CLINICAL TRIAL: NCT06954181
Title: Quantification of Diclofenac 2.32% (Voltaren) in Rinse Water After Different Application Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 300272
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Voltaren® Schmerzgel forte; 2.32% Applied Without Applicator (Method 1) (Experimental): Participants will apply the test product (Voltaren® Schmerzgel forte; 2.32%) topically on the assigned test area (left or right elbow, depending on the handedness of the participant) using 3 different methods, once on Days 1, 3 and 5 as per crossover assignment. There will be a washout period of at least 2 days between each method. Method 1: Participants will apply the test product on the assigned test area with one hand by gently massaging in for 60 seconds and will wash their hands and 5 minutes after application, will wash the test area according to the washing procedure on Days 1, 3 and 5 as per crossover assignment. The water of each washing step will be collected separately.
  Interventions: Drug: Voltaren® Schmerzgel forte; 2.32% (Test Product)
- Voltaren® Schmerzgel forte; 2.32% Applied With Applicator (Method 2) (Experimental): Participants will apply the test product (Voltaren® Schmerzgel forte; 2.32%) topically on the assigned test area (left or right elbow, depending on the handedness of the participant) using 3 different methods, once on Days 1, 3 and 5 as per crossover assignment. There will be a washout period of at least 2 days between each method. Method 2: Participants will apply the test product on the assigned test area with the applicator, followed by washing the test area 5 minutes after application (1st washing) and 5 minutes after 1st washing (2nd washing) on Days 1, 3 and 5 as per crossover assignment. The water of each washing step will be collected separately.
  Interventions: Drug: Voltaren® Schmerzgel forte; 2.32% (Test Product)
- Voltaren® Schmerzgel forte; 2.32% Applied With Applicator (Method 3) (Experimental): Participants will apply the test product (Voltaren® Schmerzgel forte; 2.32%) topically on the assigned test area (left or right elbow, depending on the handedness of the participant) using 3 different methods, once on Days 1, 3 and 5 as per crossover assignment. There will be a washout period of at least 2 days between each method. Method 3: Participants will apply the test product on the assigned test area with the applicator followed by wiping the test area with a paper towel and washing the test area and hands according to the washing procedure after 5 minutes of application on Days 1, 3 and 5 as per crossover assignment. The water of the washing step will be collected.
  Interventions: Drug: Voltaren® Schmerzgel forte; 2.32% (Test Product)

INTERVENTIONS:
Drug: Voltaren® Schmerzgel forte; 2.32% (Test Product) — Voltaren® Schmerzgel forte; 2.32% containing 2.32% Diclofenac-N-Ethylethanamin.

SUMMARY:
The purpose of this study is to quantify the amount of diclofenac in rinse water after application of the test product (Voltaren® Schmerzgel forte; 2.32 percent [%]) containing 2.32% Diclofenac-N-Ethylethanamin either by hand or using an applicator and subsequent washing and/or wiping.

DETAILED DESCRIPTION:
This will be an exploratory, open label, crossover study. Participants with healthy skin on the elbows and hands will be enrolled. The amount of diclofenac in rinse water after application of the test product (Voltaren® Schmerzgel forte; 2.32%) containing 2.32% Diclofenac-N-Ethylethanamin will be assessed after three different washing methods, with and without use of an applicator in a crossover design. There will be a wash-out period of at least 2 days in between each method. Approximately 40 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Willingness to actively participate in the study and to come to the scheduled visits.
* Female and/or male.
* From 18 to 70 years of age.

Exclusion Criteria:

* Female participants: Pregnancy or lactation.
* Drug addicts, alcoholics.
* Acquired immunodeficiency syndrome (AIDS), human immunodeficiency virus (HIV)-positive or infectious hepatitis.
* Conditions which exclude a participation or might influence the test reaction/evaluation.
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area.
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years.
* A previous allergic reaction, sensitivity or intolerance to diclofenac or any of the other ingredients in Voltaren® Schmerzgel forte.
* Participants in whom asthma, angioedema, urticaria or acute rhinitis are precipitated by acetyl salicylic acid or other non-steroidal anti-inflammatory drugs (example, ibuprofen, naproxen et cetera).
* Documented allergies to cosmetic products.
* Active skin disease at the test area.
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, et cetera, at the test area that could influence the investigation.
* Any topical medication at the test area within the last 3 days prior to the start of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Concentration of Voltaren® Schmerzgel forte; 2.32% (Diclofenac) in Water (Milligrams per Liter [mg/L]) | Day 1, Day 3 and Day 5
  The concentration of diclofenac in rinse water samples (mg/L) collected after application of the test product (Voltaren® Schmerzgel forte; 2.32%) either by hand or using an applicator and subsequent washing will be determined with High-performance liquid chromatography (HPLC).
Amount of Test Product Residues by Gravimetrical Measurements (Milligrams [mg]) | Day 1, Day 3 and Day 5
  Test product (Voltaren® Schmerzgel forte; 2.32%) residues will be collected using Method 3 (application of the test product using an applicator and subsequent wiping with a paper towel and washing). The paper towels will be weighed before and after application. The amount of test product residues (mg) in paper towel will be determined using gravimetrical measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.